CLINICAL TRIAL: NCT07068451
Title: A Prospective Randomized Study Comparing Greater Occipital Nerve Block Alone Versus Dual Nerve Blockade in the Management of Cervicogenic Headache and Occipital Neuralgia
Brief Title: Greater Occipital Nerve Block Alone Versus Dual Nerve Block in Cervicogenic Headache and Occipital Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University Hospital (Other)
Responsible Party: Principal Investigator, Ali Hammed, Dr, Tishreen University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/2020-31
Record Dates: First submitted 2025-06-26; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ervicogenic Headache (CEH); Occipital Neuralgia (ON)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GONB Alone (Experimental): Patients received a single injection of 1 mL of 2% lidocaine at the greater occipital nerve using a landmark-guided technique.
  Interventions: Procedure: Greater Occipital Nerve Block (GONB)
- GONB + LONB (Dual Block) (Experimental): Patients receive two injections of 1 mL of 2% lidocaine each at the greater and lesser occipital nerves using a landmark-guided technique.
  Interventions: Procedure: Combined Greater and Lesser Occipital Nerve Block (GONB + LONB)

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block (GONB) — A landmark-guided injection of 1 mL of 2% lidocaine administered at the anatomical location of the greater occipital nerve (GON) to treat cervicogenic headache and occipital neuralgia. Performed without corticosteroids or imaging guidance.
  Other Names: Drug: Lidocaine 2%
  Arms: GONB Alone
Procedure: Combined Greater and Lesser Occipital Nerve Block (GONB + LONB) — Two landmark-guided injections of 1 mL of 2% lidocaine each at the anatomical locations of the greater and lesser occipital nerves. Performed without corticosteroids or imaging, targeting broader nerve involvement in cervicogenic headache and occipital neuralgia.
  Other Names: Drug: Lidocaine 2%
  Arms: GONB + LONB (Dual Block)

SUMMARY:
This study looked at two types of nerve block injections used to treat people with cervicogenic headache (CEH) and occipital neuralgia (ON)-two painful conditions that often cause pain at the back of the head and neck. The injections target nerves in the upper neck that may be causing the pain.

The researchers compared:

One nerve injection (greater occipital nerve block, or GONB), versus

Two nerve injections (GONB plus lesser occipital nerve block, or LONB).

ELIGIBILITY:
Adults aged 18 to 65 years

Clinical diagnosis of cervicogenic headache (CEH) and/or occipital neuralgia (ON) according to ICHD-3 criteria

Pain duration of more than 3 months

Pain localized to the occipital region, consistent with the distribution of the greater and/or lesser occipital nerves

Inadequate response to conservative therapy (e.g., analgesics, physiotherapy)

Willingness to participate and provide written informed consent

Exclusion Criteria:

Previous nerve block or other interventional procedures for headache

Use of systemic corticosteroids within the past 3 months

Known allergy to lidocaine or other amide-type local anesthetics

Evidence of secondary causes of headache on imaging (e.g., tumor, infection)

Pregnancy or breastfeeding

Active infection at the injection site

Coagulopathy or use of anticoagulant therapy

Significant psychiatric or neurological comorbidities interfering with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity measured by the Visual Analog Scale (VAS) | Baseline, 24 hours, 3 weeks, and 3 months post-intervention
  ain intensity was assessed using a 10-point Visual Analog Scale (VAS), with 0 indicating no pain and 10 indicating the worst pain imaginable. VAS scores were recorded at baseline and follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Latakia, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29368949/